CLINICAL TRIAL: NCT01806506
Title: Randomized Clinical Trial Comparing Laparoscopic Sleeve Gastrectomy and Gastric Bypass for Morbid Obesity and Underlying Metabolic and Hormonal Abnormalities
Brief Title: Randomized Comparison of Laparoscopic Sleeve Gastrectomy and Gastric Bypass for Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBN N N403 3882 33
Record Dates: First submitted 2013-01-31; First posted 2013-03-07 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2013-01

CONDITIONS: Morbid Obesity; Metabolic Syndrome X; Diabetes Mellitus; Dyslipidemia; Hypertension
Keywords: Bariatric surgery; Gastric bypass; Sleeve gastrectomy; Weight loss; Lipoproteins; Insulin resistance; Incretins; Quality of life
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome; Diabetes Mellitus; Dyslipidemias; Hypertension; Weight Loss; Insulin Resistance | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic sleeve gastrectomy (Experimental): The group of morbidly obese patients assigned to laparoscopic sleeve gastrectomy.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- Roux-en-Y Gastric Bypass (Experimental): The group of morbidly obese patients assigned to Roux-en-Y gastric bypass.
  Interventions: Procedure: Roux-en-Y Gastric Bypass

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Laparoscopic sleeve gastrectomy (LSG) is a restrictive bariatric procedure. LSG involves resection of a large part of the body and fundus of the stomach starting from the antrum up to the angle of His. The remaining part of the stomach (the gastric sleeve) is calibrated with a 36 French bougie.
  Arms: Laparoscopic sleeve gastrectomy
Procedure: Roux-en-Y Gastric Bypass — Roux-en-Y gastric bypass (RYGB) is an intermediate (restrictive and malabsorptive) operation. RYGB involves creation of a 15-20 mL gastric pouch that is anastomosed to a 100cm Roux limb created at 100cm from the ligament of Treitz.
  Arms: Roux-en-Y Gastric Bypass

SUMMARY:
Bariatric surgery is the most effective treatment for morbid obesity. Roux-en-Y gastric bypass (RYGB) is a bariatric procedure with known safety and effectiveness. Laparoscopic sleeve gastrectomy (LSG) is a newer procedure gaining popularity. The aim of the study is to compare outcomes of these two surgical methods in terms of weight loss, improvement of common comorbidities of obesity and influence on metabolic and hormonal status.

DETAILED DESCRIPTION:
Authors of the study believe that a more detailed head-to-head comparison of RYGB and LSG is necessary. The former method is the established "gold standard" procedure with good outcomes reported in many studies. However it is much more complex and the learning curve is longer. The latter method was introduced as an initial procedure in superobese patients because of its relative simplicity. It produced good outcomes in this population of superobese patients and surgeons in some centers started to use it as a primary bariatric procedure. RYGB is a restrictive and partially malabsorptive procedure and it is believed to have additional benefits in patients with metabolic disorders such as type 2 diabetes and dyslipidemia. Purely restrictive procedures such as LSG are theoretically less beneficial in this group of patients. In the present study authors will look at weight loss as well as improvement in comorbidities and several biochemical parameters and indices to assess also metabolic action of these two procedures.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥40 kg/m2
* BMI≥35 kg/m2 with at least one comorbidity associated with obesity

Exclusion Criteria:

* BMI > 60 kg/m2
* poorly controlled significant medical or psychiatric disorders
* active alcohol or substance abuse
* active duodenal/gastric ulcer disease
* difficult to treat gastro-esophageal reflux disease with a large hiatal hernia
* previous major gastrointestinal surgery
* diagnosed or suspected malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2008-11; Primary Completion 2012-03 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Paluszkiewicz, Prof. MD,PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of General, Transplant and Liver Surgery, Public Central Teaching Hospital, Medical University of Warsaaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalinowski P, Paluszkiewicz R, Ziarkiewicz-Wroblewska B, Wroblewski T, Remiszewski P, Grodzicki M, Krawczyk M. Liver Function in Patients With Nonalcoholic Fatty Liver Disease Randomized to Roux-en-Y Gastric Bypass Versus Sleeve Gastrectomy: A Secondary Analysis of a Randomized Clinical Trial. Ann Surg. 2017 Nov;266(5):738-745. doi: 10.1097/SLA.0000000000002397. PMID 28767558
- See also: Medical University of Warsaw web site — http://www.wum.edu.pl
- See also: Chair and Department of General Transplant and Liver Surgery, Medical University of Warsaw — https://hepaclin.wum.edu.pl/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from the population of patients referred for bariatric consultation to the outpatient clinic of the Department of General, Transplant and Liver Surgery, Medical University of Warsaw, Poland. The recruitment started in November 2008 and finished when the planned number of patients had been recruited for the study.
Pre-assignment Details: Eighty six patients meeting the general criteria for bariatric surgery were evaluated for eligibility for the study. Six patients did not meet eligibility criteria (age > 60 years in 5 patients, suspicion of malignancy in 1 patient) and 8 patients decided not to participate in the study.
Period: Overall Study
Arm/Group | Laparoscopic Sleeve Gastrectomy | Roux-en-Y Gastric Bypass
Started | 36 | 36
1 Month | 36 | 36
3 Months | 35 (1 patient (reason - lost contact)) | 36
6 Months | 34 (1 patient (reason - lost contact)) | 36
9 Months | 34 | 35 (1 patient (reason - lost contact))
Completed | 34 | 35
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Sleeve Gastrectomy | Roux-en-Y Gastric Bypass | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (10.6) | 43.9 (10.8) | 44.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  Poland | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Excess Weight Loss From Baseline
Description: Weight loss measured as a percentage of excess weight lost is one of the most commonly used and accepted outcome measure in clinical trials evaluating bariatric surgery.
Time Frame: 12 months after surgery
Measure: Mean (Standard Deviation); unit: percentage of EWL
Arm/Group | Laparoscopic Sleeve Gastrectomy | Roux-en-Y Gastric Bypass
Number analyzed (Participants) | 36 | 36
percentage of EWL | 67.8 (19.3) | 64.2 (18.5)

2. Secondary Outcome: Number of Patients With Complications
Description: Complications are defined as any negative deviation from the normal postoperative course. Complications of bariatric surgery include but are not limited to: gastrointestinal leak, intrabdominal bleeding, gastrointestinal bleeding, gastrointestinal stricture, gastrointestinal fistula, marginal ulceration, internal hernia, bowel obstruction, deep vein thrombosis, pulmonary embolism, wound infection, seroma, fascial dehiscence, abdominal hernia, gallstone formation, dehydration, nutritional deficiencies
Time Frame: 12 months after surgery
Reporting Status: Not Posted

3. Secondary Outcome: Comorbidities Prevalence Changes
Description: Number of patients with comorbidities such as: type 2 diabetes mellitus, arterial hypertension, dyslipidemia, obstructive sleep apnea, degenerative arthritis, gallbladder disease, gastro-esophageal reflux disease.
Time Frame: Evaluation at baseline and 1, 6 and 12 months after surgery
Reporting Status: Not Posted

4. Secondary Outcome: Change in Weight From Baseline
Description: Absolute weight loss (in kilograms) is evaluated. It is one of the most commonly used and accepted outcome measures in clinical trials evaluating bariatric surgery. It is more dependent on the initial weight of a study participant.
Time Frame: Evaluation at baseline and 12 months after surgery
Reporting Status: Not Posted

5. Secondary Outcome: Change in BMI From Baseline
Description: Assessment of Body Mass Index (weight divided by height in meters squared) change from baseline.
Time Frame: Baseline and 12 months after surgery
Reporting Status: Not Posted

6. Secondary Outcome: Plasma Total Cholesterol at 12 Months
Description: Fasting plasma total cholesterol concentration in patients 12 months after surgery.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

7. Secondary Outcome: Plasma HDL at 12 Months
Description: Fasting plasma high density lipoprotein (HDL) cholesterol concentration in patients 12 months after surgery.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

8. Secondary Outcome: Plasma LDL at 12 Months
Description: Fasting plasma low density lipoprotein (LDL) cholesterol concentration in patients 12 months after surgery.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

9. Secondary Outcome: Plasma Triglycerides at 12 Months
Description: Fasting plasma triglycerides concentration in patients 12 months after surgery.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

10. Secondary Outcome: Plasma Glucose at 12 Months
Description: Fasting plasma glucose concentration in patients 12 months after surgery.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

11. Secondary Outcome: Plasma Insulin at 12 Months
Description: Fasting plasma insulin concentration in patients 12 months after surgery.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

12. Secondary Outcome: Plasma C-peptide at 12 Months
Description: Fasting plasma C-peptide concentration in patients 12 months after surgery.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

13. Secondary Outcome: HOMA Index at 12 Months
Description: Insulin resistance (IR) measured with the homeostatic model assessment (HOMA) method. In the published studies the HOMA model correlated with estimates using the reference euglycemic clamp method. The following equation is used: HOMA-IR = (fasting plasma glucose concentration [mmol/L] x fasting plasma insulin concentration [miliunits/L])/22.5
Time Frame: 12 months after surgery
Reporting Status: Not Posted

14. Secondary Outcome: HbA1c at 12 Months
Description: The proportion of glycosylated hemoglobin (HbA1c) [%] is measured to assesses the average plasma glucose concentration and regulation.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

15. Secondary Outcome: Plasma CRP at 12 Months
Description: C-reactive protein (CRP) is used as a marker of inflammation. It may be also used in the assessment of heart disease risk.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

16. Secondary Outcome: Plasma Uric Acid at 12 Months
Description: Hyperuricemia is associated with metabolic syndrome and obesity.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

17. Secondary Outcome: Plasma Ghrelin at 12 Months
Description: Ghrelin is an appetite-stimulating hormone produced in the fundus of the stomach. Its concentration may change after some bariatric procedures.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

18. Secondary Outcome: Plasma Leptin at 12 Months
Description: Leptin is one of the adipose-derived hormones that causes inhibition of appetite. Elevated leptin levels are associated with obesity, inflammation, metabolic syndrome and cardiovascular disease. Weight loss leads to a decline in leptin concentrations.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

19. Secondary Outcome: Plasma Glucagon at 12 Months
Description: Glucagon is synthesized and secreted from alpha cells of the pancreas. It leads to elevation of the plasma glucose.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

20. Secondary Outcome: Plasma IGF-1 at 12 Months
Description: Insulin like growth factor 1 (IGF-1) is similar in structure to insulin. It has anabolic effects. Its levels may be related to BMI and level of nutrition.
Time Frame: 12 months after surgery
Reporting Status: Not Posted

21. Secondary Outcome: AST Level
Time Frame: 12 months
Reporting Status: Not Posted

22. Secondary Outcome: ALT Level
Time Frame: 12 months
Reporting Status: Not Posted

23. Secondary Outcome: INR
Time Frame: 12 months
Reporting Status: Not Posted

24. Secondary Outcome: Albumin Level
Time Frame: 12 months
Reporting Status: Not Posted

25. Secondary Outcome: GGT Level
Time Frame: 12 months
Reporting Status: Not Posted

26. Secondary Outcome: ALP Level
Time Frame: 12 months
Reporting Status: Not Posted

27. Secondary Outcome: LDH Level
Time Frame: 12 months
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Quality of Life Questionnaire Score
Description: Quality of life questionnaire score at 12 months(WHO-Bref Quality of Life questionnaire)
Time Frame: 12 months after surgery
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Pulmonary Function Changes at 12 Months
Description: Spirometry and plethysmography results are used to assess pulmonary function before and after surgery.
Time Frame: Baseline and 12 months from surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Laparoscopic Sleeve Gastrectomy | Roux-en-Y Gastric Bypass
Serious Adverse Events (participants affected / at risk) | 3/36 | 0/36
Other Adverse Events (participants affected / at risk) | 3/36 | 6/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Sleeve Gastrectomy (N=36) | Roux-en-Y Gastric Bypass (N=36)
Gastric leak (Gastrointestinal disorders) | 1 (1) | 0 (0) — Non-symptomatic gastric leak observed in a water-soluble contrast swallow study. Treated with relparoscopy and drainage with no further complications.
Bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0) — Intragastric bleeding - one case treated laparoscopically, the other required reoperation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Sleeve Gastrectomy (N=36) | Roux-en-Y Gastric Bypass (N=36)
Wound infection (Surgical and medical procedures) | 1 (1) | 2 (2)
Fluid collection (Surgical and medical procedures) | 2 (2) | 4 (4) — Seroma

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No